CLINICAL TRIAL: NCT01675284
Title: A Phase I, Prospective, Randomized, Open Label, Observer-Blind, Single Center Study to Evaluate the Safety, Reactogenicity and Immunogenicity of an Inactivated H5N1 Influenza Vaccine Produced in Madin-Darby Canine Kidney (MDCK) Cells
Brief Title: A Phase I Study to Evaluate the Safety, Reactogenicity, and Humoral Immune Responses to an Inactivated H5N1 Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medigen Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CT-AI-11
Record Dates: First submitted 2012-08-22; First posted 2012-08-29 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Bird Flu; Avian Influenza; Influenza A(H5N1)
Keywords: Avian Influenza; Influenza A Virus Subtype H5N1; Inactivated H5N1 Influenza Virion Vaccine; Phase I; Preventive H5N1 vaccination
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dosage AT-301 (Experimental): 7.5 µg hemagglutinin (HA)
  Interventions: Biological: AT-301
- Middle Dosage AT-301 (Experimental): 15 µg hemagglutinin (HA)
  Interventions: Biological: AT-301
- High Dosage AT-301 (Experimental): 30 µg hemagglutinin (HA)
  Interventions: Biological: AT-301

INTERVENTIONS:
Biological: AT-301 — Inactivated H5N1 Influenza Virion Vaccine

SUMMARY:
The focus of this study is to evaluate the safety, reactogenicity and humoral immune responses of the study vaccine when administered at the dose of 7.5 µg HA, 15 µg HA, or 30 µg HA to human subjects.

DETAILED DESCRIPTION:
Since 1997, avian H5N1 influenza in Southeast Asia has caused several human infections and has a high mortality rate. Experts warn that the next influenza pandemic is imminent and could be severe and prevention and control will depend on the rapid production and worldwide distribution of specific pandemic influenza candidate vaccines. An H5N1 influenza vaccine was successfully produced from whole virus grown in MDCK (Madin-Darby canine kidney) cells. These purified inactivated vaccine antigens were safe and could induce immune responses in animal studies. Moreover, when formulated in aluminum phosphate a stronger response was generated even at low doses in animals (Chong et al., 2008; Hu et al., 2008). However, further investigations are necessary before their human safety and immunogenicity can be established. This human phase I clinical study, therefore, evaluates the safety and immunogenicity of adjuvanted H5N1 virion influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥20 and ≤60 years of age
* In good health as determined by medical history, physical examination, and clinical judgment of the investigator
* Willing and able to comply with all required study visits and follow-up required by this protocol
* Must provide written informed consent

Exclusion Criteria:

* Known or potential exposure to avian influenza virus or any H5N1 HA antigen vaccine
* Had any influenza vaccine within 6 months
* Administered with any vaccine within 30 days
* A history of hypersensitivity to vaccines or inflammatory or degenerative neurological disease
* Receiving chronic administration of immunosuppressants or other immune-modifying drugs within 6 months
* Known HIV, hepatitis B (HBsAg) or hepatitis C seropositivity
* Any medical illness including clinically significant acute pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests
* Receiving immunoglobulins and/or any blood products within the three months
* Acute disease at the time of enrolment
* Psychiatric, addictive, or any disorder, which may compromise the ability to give a truly informed consent for participation of this study or adequate compliance
* Breast feeding or pregnant women

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Signs and symptoms solicited by vaccination | A 7-day follow-up period after each vaccine administration
  Percentage, intensity, and relationship to vaccination of solicited local and general signs and symptoms during a 7-day follow-up period (i.e. day of vaccination and 6 subsequent days) after each administered vaccine.
Signs and symptoms unsolicited by vaccination | A 21-day follow-up period after each vaccine administration
  Percentage, intensity, and relationship to vaccination of unsolicited local and general signs and symptoms during a 21-day follow-up period (i.e. day of vaccination and 20 subsequent days) after each administered vaccine.
Occurrence of adverse events and serious adverse events | Up to 180 days after the first vaccine administration
  Occurrence of overall adverse events and serious adverse events up to 180 days after the first administered vaccine.

SECONDARY OUTCOMES:
Serum antibody titers to H5N1 virus | Day 0
  Serum anti-HA antibody titers and neutralizing antibody titers.
Serum antibody titers to H5N1 virus | Day 21
  Serum anti-HA antibody titers and neutralizing antibody titers.
Serum antibody titers to H5N1 virus | Day 42
  Serum anti-HA antibody titers and neutralizing antibody titers.

CONTACTS AND LOCATIONS:
Overall Officials: Pan-Chyr Yang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Cheng A, Hsieh SM, Pan SC, Li YH, Hsieh EF, Lee HC, Lin TW, Lai KL, Chen C, Shi-Chung Chang S, Chang SC. The safety and immunogenicity of a cell-derived adjuvanted H5N1 vaccine - A phase I randomized clinical trial. J Microbiol Immunol Infect. 2019 Oct;52(5):685-692. doi: 10.1016/j.jmii.2019.03.009. Epub 2019 May 18. PMID 31255574